CLINICAL TRIAL: NCT03896893
Title: Impact of 1% Chlorhexidine Gluconate and/or Emollient on Neonatal Bacterial Colonization Dynamics
Brief Title: Neonatal Bacterial Colonization Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Stellenbosch (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Angela Dramowski, Associate Professor, University of Stellenbosch
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: N18/07/068; 5K43TW010682 (NIH)
Record Dates: First submitted 2019-03-25; First posted 2019-04-01 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Neonatal SEPSIS; Prematurity; Very Low Birth Weight Baby; Bloodstream Infection
MeSH Terms: conditions — Neonatal Sepsis; Premature Birth; Sepsis | interventions — Emollients

STUDY DESIGN:
Intervention Model Description: Enrolled babies will be sequentially recruited to one of 4 study arms (see below).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard of Care (No Intervention): Routine bathing and skin care as per hospital practice
- 1% chlorhexidine gluconate (CHG) (Experimental): 1% aqueous CHG applied from the neck down with cotton swabs daily on weekdays (total of 8 days CHG application)
  Interventions: Other: Skin antisepsis
- Emollient therapy (Experimental): Aquaphor skin cream applied from the neck down daily on weekdays (total of 8 days emollient application)
  Interventions: Other: Emollient
- 1% CHG plus emollient therapy (Experimental): 1% aqueous CHG applied from the neck down with cotton swabs daily on weekdays followed immediately by Aquaphor skin cream (total of 8 days CHG application plus emollient application)
  Interventions: Other: Skin antisepsis; Other: Emollient

INTERVENTIONS:
Other: Skin antisepsis — 1% aqueous chlorhexidine gluconate
  Arms: 1% CHG plus emollient therapy; 1% chlorhexidine gluconate (CHG)
Other: Emollient — Aquaphor skin cream
  Arms: 1% CHG plus emollient therapy; Emollient therapy

SUMMARY:
This study will evaluate the effect of skin antisepsis and/or emollient therapy on bacterial colonization dynamics in very low birth weight, hospitalized infants. Bacterial swabs from 5 body sites will be collected at baseline, day 3, day 8 and day 13 following study arm assignment. Study outcomes include changes in bacterial colony counts, burden of gram-negative and gram-positive pathogens and overall skin score.

DETAILED DESCRIPTION:
Despite substantial global decline in childhood mortality rates, equivalent progress in neonatal mortality reduction has not been achieved. Severe bacterial infection affects approximately 6.9 million neonates and causes an estimated 750 000 deaths in low-middle income countries (LMIC) annually. The neonatal period extends from birth to 28 days of life, although neonatal hospitalization episodes (and therefore infection risk) are often substantially prolonged in preterm infants. In South Africa, infections account for 13.8% of neonatal mortality (following prematurity and intrapartum hypoxia). The South African Perinatal Problem Identification Programme (PPIP) cites nosocomial infection as the second most prevalent avoidable factor in neonatal deaths. Developing new approaches to prevent infection in hospitalized and preterm newborns in LMIC is key to achieving the Sustainable Development targets for under-five child survival.

The risk for hospital-onset sepsis in African neonates is disproportionately high and influenced by many factors including: high rates of prematurity and low birth weight; increasing in-hospital births, understaffing of maternity and neonatal services and limited implementation of infection prevention practices. Of infections among hospitalized neonates in high-income settings, hospital-acquired bloodstream infections (HA-BSI) predominate, accounting for 57% of infections. Research addressing the problem of hospital-onset neonatal infection should therefore focus on BSI prevention. A key target for sepsis reduction is prevention of intrapartum and post-delivery acquisition of bacterial colonization. Although the pathogenesis of bacterial colonization preceding invasive infection is well-accepted, there is limited data describing neonatal bacterial colonization dynamics in low-resource settings. Full characterization of timing, source and route of bacterial acquisition, flora/pathogen distribution, balance and changes over time is needed to identify all potential targets for neonatal BSI prevention.

Emollient therapy and reduction of pathogen colonization through skin antisepsis, are potentially useful targets for reducing risk of hospital-acquired BSI in neonates. Emollients (oils, creams and ointments) have been applied daily or bi-daily in neonatal research and routine practice settings, to promote skin integrity in preterm infants <37 weeks' gestation. The postulated mechanism of effect is improved skin barrier function and promotion of normal flora colonization, which may prevent pathogen ingress and subsequent invasive infection. A 2016 Cochrane review of emollient therapy for sepsis prevention in preterm infants found no evidence of reduced mortality or bloodstream infection rates, but the authors concluded that further studies in low-resource settings were warranted.

Chlorhexidine gluconate (CHG) is a bisbiguanide molecule with broad-spectrum antiseptic activity producing membrane disruption through increased cell permeability and bacterial lysis. Efficacy and safety of daily CHG bathing to prevent pediatric bacteremia was established in a multicenter, cluster-randomized trial for infants >2 months in intensive care (ICU) using 2% CHG-impregnated cloths. Three high-quality studies of newborn CHG skin or cord cleansing showed reduced neonatal mortality and omphalitis in community-based neonates. Safety of topical CHG application for neonates has been established at concentrations ≤1%, although there is little data available on its use in premature, hospitalized neonates.

CHG skin cleansing and emollient therapy are potentially useful interventions for prevention of hospital-acquired BSI in neonates from low-resource settings. In addition, these interventions are suitable for inclusion in a neonatal sepsis prevention care bundle, should they be found to be effective, safe and feasible. In addition these interventions would be low-cost, easily scalable and potentially, a maternally-administered intervention. This study will evaluate the effect of skin antisepsis and/or emollient therapy on bacterial colonization dynamics in very low birth weight, hospitalized infants. Bacterial swabs from 5 body sites will be collected at baseline, day 3, day 8 and day 13 following study arm assignment. Study outcomes include changes in bacterial colony counts, burden of gram-negative and gram-positive pathogens and overall skin score.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight ≥1000g and ≤ 1500g (equivalent to gestational age 28 - 32 weeks)
* Day 1 or 2 or 3 of life
* Anticipated length of hospital stay > 7 days.

Exclusion Criteria:

* Birth weight <1000g or >1500g
* Mother not present, unable or unwilling to provide consent for enrolment
* Any skin condition or congenital defect that could potentially result in enhanced CHG absorption (skin blistering/bullae, congenital anomalies e.g. gastroschisis, spina bifida)
* Anticipated length of hospital stay < 7 days.

Max Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2019-03-04 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in median bacterial colony counts by body site over time | baseline, day 3, day 8 and day 13 post enrolment
Change in Gram negative pathogen burden by body site over time | baseline, day 3, day 8 and day 13 post enrolment
Change in Gram positive pathogen burden by body site over time | baseline, day 3, day 8 and day 13 post enrolment
Change in median skin condition score over time (Grading scale adapted by Darmstadt from Lane at al) | Daily from enrolment to day 13 post enrolment
  Darmstadt skin score uses a 9-point scale (calculated as the sum of points for each of 3 items: skin eythema, dryness and breakdown, with a minimum score of 1 and maximum score of 3, representing worst possible skin condition for each sub-scale, total sum of points is a minimum score of 3 and maximum score of 9 for worst possible skin condition)

SECONDARY OUTCOMES:
Incidence of laboratory-confirmed sepsis | up until day 28 of life
  pathogen identified on sterile site specimen (blood, urine, cerebrospinal fluid)
Incidence of clinically-suspected sepsis | up until day 28 of life
  culture-negative episode of infection with at least 5 days broad-spectrum antibiotic therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Tygerberg Hospital, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: Anticipated availability from first quarter 2020

REFERENCES:
- [Derived] Dramowski A, Pillay S, Bekker A, Abrahams I, Cotton MF, Coffin SE, Whitelaw AC. Impact of 1% chlorhexidine gluconate bathing and emollient application on bacterial pathogen colonization dynamics in hospitalized preterm neonates - A pilot clinical trial. EClinicalMedicine. 2021 Jun 18;37:100946. doi: 10.1016/j.eclinm.2021.100946. eCollection 2021 Jul. PMID 34195575